CLINICAL TRIAL: NCT06847724
Title: A Randomized, Double-blind, Parallel-group Study to Compare the Pharmacokinetics, Efficacy, Pharmacodynamics, Safety, and Immunogenicity of CYB704 (Proposed Ocrelizumab Biosimilar) and Ocrevus® in Participants With Relapsing Multiple Sclerosis (RMS) [STRIVE-MS].
Brief Title: Comparative PK, PD, Efficacy, and Safety Assessment of the Proposed Ocrelizumab Biosimilar CYB704 and Ocrevus in Participants With Relapsing Multiple Sclerosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCYB704A12301
Record Dates: First submitted 2025-02-19; First posted 2025-02-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CYB704 (Experimental): Drug: CYB704 (Ocrelizumab) Patients will be dosed 300 mg on day 1 and day 15. Subsequent dose of 600 mg will be administered 24 weeks after the initial dose.
  Interventions: Biological: CYB704
- Ocrevus-US/Ocrevus-EU (Active Comparator): Drug: Ocrevus-US/Ocrevus-EU Patients will be dosed 300 mg on day 1 and day 15 with Ocrevus-US. Subsequent dose of 600 mg Ocrevus-EU will be administered 24 weeks after the initial dose.
  Interventions: Biological: Ocrevus-EU; Biological: Ocrevus-US

INTERVENTIONS:
Biological: CYB704 — Intravenous Infusion
  Other Names: Ocrelizumab
  Arms: CYB704
Biological: Ocrevus-EU — Intravenous Infusion
  Other Names: Ocrelizumab
  Arms: Ocrevus-US/Ocrevus-EU
Biological: Ocrevus-US — Intravenous Infusion
  Other Names: Ocrelizumab
  Arms: Ocrevus-US/Ocrevus-EU

SUMMARY:
The goal of this clinical trial is to learn if drug CYB704, a proposed biosimilar to Ocrevus, works to treat multiple sclerosis in the same way as the reference product Ocrevus(R).

The main questions it aims to answer are:

* Is CYB704 distributed in the body in the same way as the reference product (demonstration of pharmacokinetic (PK) similarity)?
* Does have CYB704 the same treatment effect and side effects as the reference product?

Researchers will compare CYB704 to a Ocrevus (Ocrevus-US and Ocrevus-EU). Participants will:

* Take drug CYB704 or Ocrevus (Ocrevus-US and Ocrevus-EU)
* Visit the clinic for at least 15 treatment visits, checkups and tests
* Will undergo regular magnetic resonance imaging (MRI) examinations

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RMS (relapsing remitting multiple sclerosis (MS) or active secondary progressive MS)
* Evidence of recent disease activity as defined in study protocol
* Expanded Disability Status scale score of 0 to 5.5 (inclusive) at screening
* Neurological stability (no new signs or symptoms referable to Central Nervous System (CNS) within 30 days before both screening and first study treatment

Exclusion Criteria:

* Diagnosis of primary progressive MS
* Disease duration of more than 10 years in participants with an Expanded Disability Status Scale (EDSS) ≤2.0 at screening
* Inability to complete an MRI or contraindication to gadolinium administration
* History of allergic or anaphylactic reactions to ocrelizumab or one of the premedications (methylprednisolone or equivalent corticosteroid, antihistamine, antipyretic)
* Pregnant participants
* Current or history of medical conditions as outlined in the study protocol
* Prohibited medications (current and history) as outlined in the study protocol
* Abnormal laboratory blood values as outlined in the study protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-10-14 (Estimated); Study Completion 2029-10-14 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration time curve | Week 1 - 3, week 3 - 25
  Demonstrate similar PK between Ocrevus and CYB704

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Week 1 - 25
  Compare PK between Ocrevus and CYB704
Peak Plasma Concentration (Cmax) | Day 1 and Day 15
  Demonstrate similar PK between Ocrevus and CYB704
CD19+ B-cell count | Up to 48 weeks
  Compare PD between Ocrevus and CYB704
Number of new T1 GdE lesions on brain MRI scans | Up to 48 weeks
  Compare efficacy between Ocrevus and CYB704
Number of T1 GdE lesions | Up to 48 weeks
  Compare efficacy between Ocrevus and CYB704
Number of new/enlarging T2 lesions | Up to 48 weeks
  Compare efficacy between Ocrevus and CYB704
Number of combined unique active lesions | Up to 48 weeks
  Compare efficacy between Ocrevus and CYB704
Annualized Relapse Rate | Up to 48 weeks
  Compare efficacy between Ocrevus and CYB704
Treatment emergent Adverse Events and Serious Adverse Events | Up to 48 weeks
  Compare safety between Ocrevus and CYB704
Rate of patients with anti-drug antibodies | Up to 48 weeks
  Compare immunogenicity between Ocrevus and CYB704

CONTACTS AND LOCATIONS:
Locations (38):
- United States (2):
  - Sandoz Investigational Site, Maitland, Florida
  - Sandoz Investigational Site, Ormond Beach, Florida
- Bosnia and Herzegovina (4):
  - Sandoz Investigational Site, Banja Luka
  - Sandoz Investigational Site, Bihać
  - Sandoz Investigational Site 2, Sarajevo
  - Sandoz Investigational Site, Sarajevo
- Bulgaria (8):
  - Sandoz Investigational Site, Pleven
  - Sandoz Investigational Site 2, Plovdiv
  - Sandoz Investigational Site, Plovdiv
  - Sandoz Investigational Site 2, Sofia
  - Sandoz Investigational Site 3, Sofia
  - Sandoz Investigational Site 4, Sofia
  - Sandoz Investigational Site 5, Sofia
  - Sandoz Investigational Site, Sofia
- Croatia (2):
  - Sandoz Investigational Site, Varaždin
  - Sandoz Investigational Site, Zagreb
- Georgia (8):
  - Sandoz Investigational Site, Rustavi
  - Sandoz Investigational Site 2, Tbilisi
  - Sandoz Investigational Site 3, Tbilisi
  - Sandoz Investigational Site 4, Tbilisi
  - Sandoz Investigational Site 5, Tbilisi
  - Sandoz Investigational Site 6, Tbilisi
  - Sandoz Investigational Site 7, Tbilisi
  - Sandoz Investigational Site, Tbilisi
- North Macedonia (2):
  - Sandoz Investigational Site, Shtip
  - Sandoz Investigational Site, Skopje
- Poland (10):
  - Sandoz Investigational Site, Bydgoszcz
  - Sandoz Investigational Site 2, Katowice
  - Sandoz Investigational Site, Katowice
  - Sandoz Investigational Site, Lodz
  - Sandoz Investigational Site, Nowa Sól
  - Sandoz Investigational Site 2, Poznan
  - Sandoz Investigational Site, Poznan
  - Sandoz Investigational Site, Szczecin
  - Sandoz Investigational Site, Warsaw
  - Sandoz Investigational Site, Zabrze
- Serbia (2):
  - Sandoz Investigational Site, Belgrade
  - Sandoz Investigational Site, Niš

IPD SHARING:
Plan to Share IPD: No